CLINICAL TRIAL: NCT00391716
Title: Gabapentin Treatment of Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, PI, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAAMAS014028; R37AA014028 (NIH)
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Alcoholism; Alcohol Dependence
Keywords: Alcohol; Alcohol treatment; Alcoholism; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Gabapentin; Behavior Therapy; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- gabapentin 900mg daily (Experimental): 900mg gabapentin daily for 12 weeks and weekly concomitant manualized behavioral counseling for 12 weeks.
  Interventions: Drug: Gabapentin 900mg; Behavioral: behavioral counseling
- gabapentin 1800mg daily (Experimental): 1800 mg gabapentin daily for 12 weeks and weekly concomitant manualized behavioral counseling for 12 weeks
  Interventions: Behavioral: behavioral counseling; Drug: gabapentin 1800mg
- placebo daily (Placebo Comparator): placebo capsules daily for 12 weeks and weekly concomitant manualized behavioral counseling for 12 weeks.
  Interventions: Behavioral: behavioral counseling; Drug: placebo

INTERVENTIONS:
Drug: Gabapentin 900mg — 900 mg gabapentin daily for 12 weeks
  Other Names: Neurontin
  Arms: gabapentin 900mg daily
Behavioral: behavioral counseling — The manual for standardized alcohol-related behavioral counseling was developed by Drs. Barbara Mason and Anita Goodman. The manual is available at alcoholfree.info.
  Other Names: alcoholfree.info
Drug: placebo — lactose capsule compounded to mimic gabapentin capsules
  Other Names: lactose capsule
  Arms: placebo daily
Drug: gabapentin 1800mg — 1800 mg gabapentin daily for 12 weeks
  Other Names: Neurontin
  Arms: gabapentin 1800mg daily

SUMMARY:
Gabapentin treatment for alcohol dependence

DETAILED DESCRIPTION:
This is a 12-week, double blind, placebo controlled, dose ranging study to evaluate the efficacy of gabapentin in treating outpatients with alcohol dependence. Subjects receive 900mg or 1800mg gabapentin or placebo daily for 12 weeks accompanied by weekly standardized counseling for alcohol-related behavior, with assessments of alcohol consumption, mood, sleep and alcohol-craving performed each week.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over age 18 with alcohol dependence

Exclusion Criteria:

* Currently meets Diagnostic and Statistical Manual 4 Text Revision (DSM-IV-TR) criteria for dependence on illicit substances
* Significant medical disorders that will increase potential risk or interfere with study participation
* Women with childbearing potential who are pregnant, nursing, or refuse to use a reliable method of birth control
* Treatment with an investigational drug in the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-02; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, PhD, Principal Investigator — The Scripps Research Institute Pearson Center for Alcoholism and Addiction Research
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

REFERENCES:
- [Result] Mason BJ, Quello S, Goodell V, Shadan F, Kyle M, Begovic A. Gabapentin treatment for alcohol dependence: a randomized clinical trial. JAMA Intern Med. 2014 Jan;174(1):70-7. doi: 10.1001/jamainternmed.2013.11950. PMID 24190578

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin 900mg Daily | Gabapentin 1800mg Daily | Placebo Daily
Started | 54 | 47 | 49
Completed | 27 | 28 | 30
Not Completed | 27 | 19 | 19

BASELINE CHARACTERISTICS:
Population: Sample size estimate was derived from results of a prior trial that found an odds ratio of 2.96 for complete abstinence, estimating a sample size of 150 would show a medium effect size for the difference between gabapentin and placebo in rate of complete abstinence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin 900mg Daily | Gabapentin 1800mg Daily | Placebo Daily | Total
Number analyzed (Participants) | 54 | 47 | 49 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (10.1) | 45.2 (11.3) | 46.8 (11.3) | 44.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 28 | 65
  Male | 33 | 31 | 21 | 85
Meets Criteria for DSM-IV Alcohol Dependence [Number; unit: participants] — Meets DSM-IV criteria for current Alcohol Dependence defined as three or more symptoms of dependence.
  participants | 54 | 47 | 49 | 150

OUTCOME MEASURES:

1. Primary Outcome: Drinking
Description: Rate of complete abstinence was defined as the number of participants who drank no alcohol during 12 weeks of treatment, where the denominator is the intent to treat population. Rate of heavy drinking abstinence is defined as no heavy drinking days while on study (4 or more for women, 5 or more for men).
Time Frame: 12-week
Population: All randomized subjects included in denominator for rate determination.
Measure: Number; unit: participants
Arm/Group | Gabapentin 900mg Daily | Gabapentin 1800mg Daily | Placebo Daily
Number analyzed (Participants) | 54 | 47 | 49
participants | 6 | 8 | 2
Statistical Analysis 1: Comparison: Gabapentin 900mg Daily vs Gabapentin 1800mg Daily vs Placebo Daily; The extended Mantel-Haenszel Chi-square test for linear trend assesses the relationship between ROW and COLUMN of a single contingency table, where both row (dose: 0mg, 900mg, 1800mg) and column (response (0= non-abstinent, 1=abstinent), and at least 1 variable has more than 2 levels. It specifically tests linear dose-response without need for multiple comparisons; Test type: Superiority or Other; p < 0.04, Mantel Haenszel — The numerator is the number of subjects completely abstinent and the denominator is the number of subjects randomized, within each treatment group; Extended Mantel-Haenszel Chi-square test for linear-by-linear association
Statistical Analysis 2: Comparison: Gabapentin 900mg Daily vs Gabapentin 1800mg Daily vs Placebo Daily; The extended Mantel-Haenszel Chi-square test for linear trend assesses the relationship between ROW and COLUMN of a single contingency table, where both row (dose: 0mg, 900mg, 1800mg) and column (response (0= heavy drinking, 1=no heavy drinking), and at least 1 variable has more than 2 levels. It specifically tests linear dose-response without need for multiple comparisons; Test type: Superiority or Other; p < 0.02, Mantel Haenszel — linear dose effects for rates of abstinence were assessed using the extended Mantel-Haenszel chi-square test for linear association; The numerator is the number of subjects completely abstinent and the denominator is the number of subjects randomized, within each treatment group

2. Secondary Outcome: Mood
Description: Beck Depression Inventory II consists of 21 questions assessing depression symptoms answered with scores between 0 and 3, summed for a weekly total score between 0 and 63; higher scores indicate more depression. The cumulative mean total depression scores over the 12 week study are tested by ANOVA for differences in cumulative means between treatment groups.
Time Frame: 12-week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin 900mg Daily | Gabapentin 1800mg Daily | Placebo Daily
Number analyzed (Participants) | 54 | 47 | 49
units on a scale | 5.08 (.53) | 3.62 (.44) | 5.40 (.39)
Statistical Analysis 1: Comparison: Gabapentin 900mg Daily vs Gabapentin 1800mg Daily vs Placebo Daily; Test type: Superiority or Other; p < 0.001, ANOVA — Cumulative means over 12 weeks

3. Secondary Outcome: Sleep
Description: The Pittsburgh Sleep Questionnaire Inventory consists of 9 questions about sleep habits which are answered on a scale of 0-3. Results are sorted into 7 sub scales re-scored 0-3, then sub scales are summed for a weekly total score between 0 and 21, with higher total scores indicating greater sleep impairment. Cumulative mean total sleep scores over the 12 weeks of study are assessed by ANOVA for differences between treatment groups.
Time Frame: 12-week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin 900mg Daily | Gabapentin 1800mg Daily | Placebo Daily
Number analyzed (Participants) | 54 | 47 | 49
units on a scale | 4.04 (.2) | 3.24 (.17) | 4.50 (.22)
Statistical Analysis 1: Comparison: Gabapentin 900mg Daily vs Gabapentin 1800mg Daily vs Placebo Daily; Test type: Superiority or Other; p < 0.001, ANOVA — Cumulative means over 12 weeks

4. Secondary Outcome: Craving
Description: Alcohol Craving Questionnaire has 12 questions about alcohol craving which are each scored 1-7, then summed for a weekly score between 7 and 84, with higher scores indicating greater craving. Cumulative mean total craving scores are tested by ANOVA for differences between treatment groups.
Time Frame: 12-week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin 900mg Daily | Gabapentin 1800mg Daily | Placebo Daily
Number analyzed (Participants) | 54 | 47 | 49
units on a scale | 33.66 (.78) | 32.31 (.82) | 34.27 (.70)
Statistical Analysis 1: Comparison: Gabapentin 900mg Daily vs Gabapentin 1800mg Daily vs Placebo Daily; Test type: Superiority or Other; p < 0.003, ANOVA — Cumulative means over 12 weeks

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Gabapentin 900mg Daily | Gabapentin 1800mg Daily | Placebo Daily
Serious Adverse Events (participants affected / at risk) | 2/54 | 0/47 | 0/49
Other Adverse Events (participants affected / at risk) | 13/54 | 9/47 | 12/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin 900mg Daily (N=54) | Gabapentin 1800mg Daily (N=47) | Placebo Daily (N=49)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Overnight Hospitalization (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin 900mg Daily (N=54) | Gabapentin 1800mg Daily (N=47) | Placebo Daily (N=49)
Fatigue (Nervous system disorders) | 13 | 9 | 12
Headache (Nervous system disorders) | 7 | 6 | 8
Insomnia (Nervous system disorders) | 10 | 6 | 11
Anxiety (Psychiatric disorders) | 2 | 5 | 6
Blurred Vision (Eye disorders) | 2 | 0 | 5
Depression (Psychiatric disorders) | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 7 | 3
Increased hunger (Metabolism and nutrition disorders) | 3 | 2 | 0
Irritability (Nervous system disorders) | 3 | 4 | 0
Cold (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2
Drowsy (Nervous system disorders) | 1 | 4 | 4
Dry Mouth (Nervous system disorders) | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes